CLINICAL TRIAL: NCT04024137
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study of ZSP1273 in Adults With Acute Uncomplicated Influenza A
Brief Title: Study of ZSP1273 in Patients With Acute Uncomplicated Influenza A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSP1273-18-02
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2019-12

CONDITIONS: Influenza A
MeSH Terms: interventions — ZSP1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZSP1273-200 mg BID (Experimental): Subjects will receive 10 doses of ZSP1273 200mg along with placebo twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5 days.
  Interventions: Drug: ZSP1273 200 mg; Drug: Placebo
- ZSP1273-400 mg BID (Experimental): Subjects will receive 10 doses of ZSP1273 400mg（200mg*2) along with placebo twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5 days.
  Interventions: Drug: ZSP1273-400 mg; Drug: Placebo
- ZSP1273-600 mg QD (Experimental): Subjects will receive 5 doses of ZSP1273 600mg （200mg *3) and 5 doses of placebo respectively for 5 days.The interval between ZSP1273 and placebo is approximately 12 hour (+/- 2) .
  Interventions: Drug: ZSP1273-600 mg; Drug: Placebo
- Placebo (Placebo Comparator): Subjects will receive 10 doses of matching placebo of ZSP1273 twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZSP1273 200 mg — 1 X 200-mg tablet taken orally
  Arms: ZSP1273-200 mg BID
Drug: Placebo — 2 tablets taken orally
  Arms: ZSP1273-200 mg BID
Drug: ZSP1273-400 mg — 2 X 200-mg tablet taken orally
  Arms: ZSP1273-400 mg BID
Drug: Placebo — 1 tablet taken orally
  Arms: ZSP1273-400 mg BID
Drug: ZSP1273-600 mg — 3 X 200-mg tablet taken orally
  Arms: ZSP1273-600 mg QD
Drug: Placebo — 3 tablets taken orally
  Arms: ZSP1273-600 mg QD
Drug: Placebo — Subjects will receive matching placebo of ZSP1273
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the antiviral effect, as measured by the time to alleviation of influenza symptoms and viral titer in nasopharyngeal secretions in adults with acute uncomplicated influenza A following administration of ZSP1273.

ELIGIBILITY:
Inclusion Criteria:

1. Males and female subjects between 18-65 years (Both inclusive).
2. Patients with a diagnosis of influenza virus A infection confirmed by all of the following:

   * Positive Rapid Antigen Test (RAT) with throat swabs;and
   * Fever≥38.0ºC (axillary) in the predose examinations;and
   * At least one of the following general systemic symptoms and respiratory symptoms respectively associated with influenza are present with a severity of moderate or greater:

     * General systemic symptoms:Headache,Feverishness or chills,Muscle or joint pain,Fatigue;
     * Respiratory symptoms:Cough,Sore throat,Nasal congestion.
3. The time interval between the onset of symptoms and the enrollment is≤48 hours. The onset of symptoms is defined as:

   * Time of the first increase in body temperature(axillary temperature≥38.0ºC),or
   * Time when the patient experiences at least one general or respiratory symptom.
4. Subjects who agree to use an appropriate method of contraception during the study and up to 6 months after drug withdrawal.
5. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.

Exclusion Criteria:

1. Known hypersensitivity and/or allergy to some drugs and food,especially for the composition that is similar to ZSP1273;
2. Dysphagia or any medical history in gastrointestinal that interferes with the absorption of drugs.
3. Use of the following medications within 7 days prior to screening:

   * Influenza antiviral medication:oseltamivir,peramivir,famivir,abidol,amantadine or rimantadine.
   * Chinese patent medicine or herbal medicine with antiviral effect.
4. Patients who have received influenza vaccine within 6 months prior to enrollment.
5. Presence of clinically significant abnormalities in ECG .
6. Chest X - ray examination confirmed bronchitis,pneumonia,pleural effusion or pulmonary interstitial lesions.
7. Patients who have experienced respiratory tract infection,Otitis media,nasosinusitis.
8. White blood cells(WBC)>10.0×109/L at screening.
9. Subject who produces purulent sputum or has suppurative tonsillitis.
10. Patients with severe or uncontrollable underlying diseases:blood disorders,severe chronic obstructive pulmonary disease(COPD),liver disorders(ALT or AST≥3 ULN,total bilirubin≥1.5 ULN),kidney disorders(serum creatinine>177μmol/L or 2mg/dL),chronic congestive heart failure(NYHA III-IV),mental disorders.
11. Immunodeficiency,including malignant tumor,organ or marrow transplant,human immunodeficiency virus [HIV] infection,or patients receiving immunosuppressant therapy 3 months prior to enrollment.
12. Concomitant therapy with aspirin or salicylic acid.
13. Morbid obesity(Body mass index [BMI]≥30kg/m2).
14. Known history of alcohol abuse or drug abuse.
15. Pregnancy or breastfeeding at screening and during the study.All female subjects of childbearing potential must have a negative urine pregnancy test at screening and during the trial.
16. Have received any other investigational products within 3 months prior to dosing.
17. Subjects who should not be included in the study in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of influenza symptoms in participants | Initiation of study treatment (Day 1) up to Day 15
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of symptoms was defined as the time from the start of the study treatment to the time when all 7 influenza-related symptoms were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours

SECONDARY OUTCOMES:
AUC of the log10 pharyngeal viral load | Days 6
  Area under the curve (AUC) of the log10 pharyngeal viral load is measured by viral culture and quantitative reverse transcriptase polymerase chain reaction (qRT-PCR).
Change in the total score of 7 influenza symptoms | Up to Day15
  Participants assessed the severity of seven influenza-associated symptoms(cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  The composite symptom score is the total score of the 7 influenza symptoms(Sum of symptom scores) as assessed by the participant, and ranges from 0 to 21.
Time to alleviation of each influenza symptom. | Up to Day15
  Participants assessed the severity of seven influenza-associated symptoms(cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of each symptom was defined as the time from the start of treatment to the start of the time period when the individual symptom was assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
Time to Resolution of Fever | Up to Day15
  Time to resolution of fever was defined as the time between the initiation of the study treatment and the resolution of fever. The resolution of fever was defined as the time when the participant's self-measured axillary temperature became less than 37ºC and was maintained at less than 37ºC for a duration of at least 12 hours.
Proportion of patients reporting normal temperature | Up to Day15
  Defined as the percentage of patients whose axillary temperature dropped to less than 37ºC after the initiation of study treatment.
Percentage of subjects with virus titer detected | Days 2,4, 6
  Influenza virus RNA was quantified from throat swabs.Proportion of patients positive for influenza virus titer is defined as the percentage of patients whose virus titer is not less than the lower limit of quantification among those assessed for virus titer measured by viral culture and quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) on Days 2,4, 6.
Duration of detectable virus | Days 2,4, 6
  Defined as the time from the start of treatment to the time when the titer is less than the lower limit of quantification measured by viral culture and quantitative reverse transcriptase polymerase chain reaction (qRT-PCR).
Change in virus titer | Days 2,4, 6
  Defined as the change from baseline in virus titer measured by viral culture and quantitative reverse transcriptase polymerase chain reaction (qRT-PCR).
Change in viral RNA load | Days 2,4, 6
  Defined as the change from baseline in viral RNA load measured by viral culture and quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) on Days 2, 4, 6.
Incidence of influenza-related complications | Up to Day21
  Defined as the percentage of subjects in the analysis population who experience each influenza-related complication (sinusitis, otitis media, bronchitis, and pneumonia) as an adverse event after the initiation of the study treatment.
Time to return to normal activities of daily life | Up to Day15
  Participants were asked to record their activities of daily life on a scale from 0 (worst possible health) to 10 (normal activities of daily life).
  Time to return to normal activities of daily life defined as the time between the initiation of the study treatment and the return to normal activities of daily life. The return to normal activities of daily life is defined as the time when the subject assesses his/her activities as 10.Subjects with a baseline self-rated daily activity score of 10 are not included in this analysis.
Proportion of patients with the Serological conversion of neutralizing antibody titer relative to that in Visit 1 ≥4 | Baseline and Day 21
  Defined as the protprtion of patients with a ratio of 4 or more at Visit 5 antibody titer relative to Visit 1 titer
Proportion of patients and frequency in combination use of acetaminophen. | Up to 21 days post-dose
  The proportion of patients who use acetaminophen in the duration of the study
Change in EQ-5D-5L | Baseline up to Day 15
  Defined as the change from baseline in the index value and that in EQ VAS score as calculated from the EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Dongguan people's Hospital, Dongguan, Guangdong
  - Nanfang Hospital,South Medical Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - Traditional Chinese Medicine Hospital of Guangdong Province, Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital Of Guangdong Medical University, Zhanjiang, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Sixth People's Hospital Of Zhengzhou, Zhengzhou, Henan
  - Sir Run Run Hospital Nanjing Medical University, Nanjing, Jiangsu
  - Jiujiang University Hospital, Jiujiang, Jiangxi
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - General Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital,Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Yang Z, Li Z, Zhan Y, Lin Z, Fang Z, Xu X, Lin L, Li H, Lin Z, Kang C, Liang J, Liang S, Li Y, Li S, Yang X, Ye F, Zhong N; Onradivir Trial Recruitment and Medical Monitoring Group. Safety and efficacy of onradivir in adults with acute uncomplicated influenza A infection: a multicentre, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2024 May;24(5):535-545. doi: 10.1016/S1473-3099(23)00743-0. Epub 2024 Feb 5. PMID 38330975